CLINICAL TRIAL: NCT04538742
Title: A Phase 1b/2 Multicentre, Open-label, Modular, Dose-finding and Dose-expansion Study to Explore the Safety, Tolerability, and Anti-tumour Activity of Trastuzumab Deruxtecan (T-DXd) in Combination With Other Anti-cancer Agents in Patients With HER2-positive Metastatic Breast Cancer (DESTINY-Breast07)
Brief Title: A Phase 1b/2 Study of T-DXd Combinations in HER2-positive Metastatic Breast Cancer
Acronym: DB-07
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo Company, Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D967JC00001; 2023-505309-18-00 (Registry Identifier: CTIS (EU)); 2019-004531-22 (EudraCT Number)
Record Dates: First submitted 2020-08-31; First posted 2020-09-04 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast Cancer; HER2-positive; Brain Metastases; Trastuzumab Deruxtecan; T-DXd; DS-8201a; DESTINY-Breast07; Anti-HER2 Antibody Drug Conjugate (ADC)
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — trastuzumab deruxtecan; durvalumab; Paclitaxel; pertuzumab; tucatinib

STUDY DESIGN:
Intervention Model Description: The study will consist of 2 phases: a dose escalation phase (Part 1) and a dose expansion phase (Part 2). Part 1 of each module will enroll patients with locally assessed HER2-positive advanced/MBC in second-line or later.Part 2 of each module will enroll patients with locally assessed HER2-positive breast cancer who have not received prior treatment for advanced/metastatic disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Module 1- T-DXd and Durvalumab (Experimental): T-DXd and Durvalumab
  Interventions: Drug: Trastuzumab deruxtecan; Drug: Durvalumab
- Module 2- T-DXd and Pertuzumab (Experimental): T-DXd and Pertuzumab
  Interventions: Drug: Trastuzumab deruxtecan; Drug: Pertuzumab
- Module 3- T-DXd and Paclitaxel (Experimental): T-DXd and Paclitaxel (Arm not initiated in Part 2)
  Interventions: Drug: Trastuzumab deruxtecan; Drug: Paclitaxel
- Module 4- T-DXd and Durvalumab and Paclitaxel (Experimental): T-DXd and Durvalumab and Paclitaxel (Arm not initiated in Part 1 and Part 2)
  Interventions: Drug: Trastuzumab deruxtecan; Drug: Durvalumab; Drug: Paclitaxel
- Module 0- T-DXd (Experimental): T-DXd
  Interventions: Drug: Trastuzumab deruxtecan
- Module 5 - T-DXd and Tucatanib (Experimental): T-DXd and tucatinib (Arm not initiated in Part 2)
  Interventions: Drug: Trastuzumab deruxtecan; Drug: Tucatinib
- Module 6 - T-DXd and Tucatinib (Experimental): T-DXd and tucatinib in patients with active brain metastases (Part 2 Only) (Arm not initiated)
  Interventions: Drug: Trastuzumab deruxtecan; Drug: Tucatinib
- Module 7 - T-DXd (Experimental): T-DXd monotherapy in patients with active brain metastases (Part 2 Only)
  Interventions: Drug: Trastuzumab deruxtecan

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — T-DXd: administered as an IV infusion
  Other Names: DS-8201a, T-DXd
Drug: Durvalumab — Durvalumab: administered as an IV infusion
  Other Names: MEDI4736
  Arms: Module 1- T-DXd and Durvalumab; Module 4- T-DXd and Durvalumab and Paclitaxel
Drug: Paclitaxel — Paclitaxel: administered as an IV infusion
  Arms: Module 3- T-DXd and Paclitaxel; Module 4- T-DXd and Durvalumab and Paclitaxel
Drug: Pertuzumab — Pertuzumab: administered as an IV infusion
  Arms: Module 2- T-DXd and Pertuzumab
Drug: Tucatinib — Tucatinib administered orally (tablet) twice daily
  Other Names: ONT-380
  Arms: Module 5 - T-DXd and Tucatanib; Module 6 - T-DXd and Tucatinib

SUMMARY:
DESTINY-Breast07 will investigate the safety, tolerability, and anti-tumour activity of trastuzumab deruxtecan (T-DXd) in combination with other anti-cancer agents in patients with HER2-positive Metastatic Breast Cancer

DETAILED DESCRIPTION:
This study is modular in design allowing assessment of safety, tolerability and anti-tumour activity of T-DXd in combination with other anti-cancer agents. Combination-treatment modules will have 2 parts: a dose-finding phase (Part 1), and a dose expansion phase (Part 2); the recommended Phase 2 dose (RP2D) determined in Part 1 will be used for the dose-expansion in Part 2.

The target population of interest in this study is patients with HER2-positive (as per ASCO/CAP 2018 guidelines) advanced/MBC inclusive of patients with active and stable brain metastases. Part 1 of each module will enroll patients with locally assessed HER2-positive advanced/MBC in second-line or later patients. Part 2 of each module will enroll patients with locally assessed HER2-positive breast cancer who have not received prior treatment for advanced/metastatic disease.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients must be at least 18 years of age
* Pathologically documented breast cancer that:

  1. Is advanced/unresectable (patients that can be treated with curative intent are not eligible) or metastatic
  2. HER2-positive (IHC 3+ or IHC 2+/ISH+) based on local assessment. The local HER2 result must be from a tumour sample obtained in the metastatic setting.
  3. Is documented as hormone receptor-positive (estrogen or progesterone receptor) or negative in the metastatic setting
* Patient must have adequate tumor sample from the metastatic setting for biomarker assessment
* ECOG Performance Status of 0 or 1
* Part 1

  1. Disease progression on or after the last systemic therapy prior to starting study treatment
  2. At least 1 prior treatment line in metastatic setting required.
* Part 2 (Modules 0 - 5)

  a) No prior lines of therapy for advanced/MBC allowed
* Part 2 (Module 6 and 7) a) Zero or one prior lines of therapy for advanced/MBC allowed

CNS Inclusion

* Modules 0 - 5 Patients must have no brain metastases or stable brain metastases.
* Module 6 and 7 Patients must have untreated brain metastases not needing local therapy or previously treated brain metastases that have progressed since prior local therapy

Key Exclusion Criteria:

* Uncontrolled or significant cardiovascular disease
* Active or prior documented (non-infectious) ILD/pneumonitis that required steroids, or suspected ILD/pneumonitis that cannot be ruled out by imaging at screening
* Lung-specific intercurrent clinically significant illnesses
* Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals
* Spinal cord compression or a history of leptomeningeal carcinomatosis
* Prior treatment with immune checkpoint inhibitors
* Prior treatment with an ADC containing a topoisomerase I inhibitor
* Prior treatment with tucatinib

CNS Exclusion

* Modules 0 - 5: Has untreated brain metastasis
* Module 6 and 7: Ongoing use of systemic corticosteroids for control of symptoms of brain metastases at a total daily dose of > 2 mg dexamethasone or any brain lesion thought to require immediate local therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse events (AEs)- Part 1 | Up to follow-up period, approximately 53 months
  Occurrence of AEs in Part 1 graded according to NCI CTCAE v5.0
Occurrence of serious adverse events (SAEs)- Part 1 | Up to follow-up period, approximately 53 months
  Occurrence of SAEs in Part 1 graded according to NCI CTCAE v5.0
Occurrence of adverse events (AEs)- Part 2 | Up to follow-up period, approximately 53 months
  Occurrence of AEs in Part 2 graded according to NCI CTCAE v5.0
Occurrence of serious adverse events (SAEs)- Part 2 | Up to follow-up period, approximately 53 months
  Occurrence of SAEs in Part 2 graded according to NCI CTCAE v5.0

SECONDARY OUTCOMES:
Objective Response Rate (ORR)- Part 1 and Part 2 | Until progression, assessed up to approximately 53 months
  ORR is defined as the proportion of patients who have a CR or PR, as determined by the Investigator at local site per RECIST 1.1.
Progression Free Survival (PFS)- Part 1 and Part 2 | Until progression, assessed up to approximately 53 months
  PFS is defined as time from the date of randomization until the date of progression as assessed by the Investigator at local site per RECIST 1.1, or death due to any cause.
Progression Free Survival 2 (PFS2)- Part 2 | Assessed up to approximately 53 months
  PFS2 is defined as time from the date of randomisation until the date of progression on next line treatment (the earliest of the progression event subsequent to first subsequent anticancer therapy) or death; second progression will be defined according to local standard clinical practice.
Duration of Response (DoR)- Part 2 | Until progression, assessed up to approximately 53 months
  DoR is defined as time from the date of first documented response until the date of documented progression or death in the absence of disease progression.
Overall Survival (OS)- Part 2 | Until death, assessed up to approximately 53 months
  OS is defined as time from the date of randomisation until the date of death due to any cause.
Serum Concentration of Trastuzumab Deruxtecan (T-DXd) | While on study drug up to study completion, approximately 53 months
  Determination of trastuzumab deruxtecan concentration in serum at different time points after trastuzumab deruxtecan administration
Serum Concentration of Durvalumab | While on study drug up to study completion, approximately 53 months
  Determination of durvalumab concentration in serum at different time points after administration
Serum Concentration of Pertuzumab | While on study drug up to study completion, approximately 53 months
  Determination of pertuzumab concentration in serum at different time points after administration
Plasma Concentration of Paclitaxel | While on study drug up to study completion, approximately 53 months
  Determination of paclitaxel concentration in plasma at different time points after administration
Plasma Concentration of Tucatinib | While on study drug up to study completion, approximately 53 months
  Determination of tucatinib concentration in plasma at different time points after administration
Immunogenicity of trastuzumab deruxtecan | Up to follow-up period, approximately 53 months
  Percentage of patients who develop ADA for trastuzumab deruxtecan
Immunogenicity of Durvalumab | Up to follow-up period, approximately 53 months
  Percentage of patients who develop ADA for durvalumab
Immunogenicity of Pertuzumab | Up to follow-up period, approximately 53 months
  Percentage of patients who develop ADA for pertuzumab

CONTACTS AND LOCATIONS:
Locations (52):
- United States (9):
  - Research Site, Fort Myers, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Commack, New York
  - Research Site, Harrison, New York
  - Research Site, New York, New York
  - Research Site, Columbus, Ohio
  - Research Site, Nashville, Tennessee
  - Research Site, Fort Worth, Texas
  - Research Site, Fairfax, Virginia
- Research Site, Melbourne, Australia
- Brazil (7):
  - Research Site, Barretos
  - Research Site, Belo Horizonte
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
  - Research Site, Sorocaba
- Canada (3):
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Toronto
- Research Site, Villejuif, France
- Germany (2):
  - Research Site, München
  - Research Site, Würzburg
- India (4):
  - Research Site, Delhi
  - Research Site, Gūrgaon
  - Research Site, Madurai
  - Research Site, Mumbai
- Italy (4):
  - Research Site, Bologna
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Rome
- Poland (4):
  - Research Site, Bydgoszcz
  - Research Site, Koszalin
  - Research Site, Lodz
  - Research Site, Lublin
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- South Korea (2):
  - Research Site, Busan
  - Research Site, Seoul
- Spain (4):
  - Research Site, Barcelona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Seville
- Taiwan (4):
  - Research Site, Hualien City
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan
- Turkey (Türkiye) (4):
  - Research Site, Ankara
  - Research Site, Edirne
  - Research Site, Istanbul
  - Research Site, Izmir
- Research Site, Buckhurst Hill, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Related Info — http://BreastCancerStudyLocator.com